CLINICAL TRIAL: NCT02217215
Title: Initial Study With the CNDS Advanced Cervical Scan to Recalibrate Spectral Data for Use in Future Screening Studies
Acronym: Spectral
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Guided Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: CLIN-4-CLP_0
Record Dates: First submitted 2014-08-05; First posted 2014-08-15 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-08

CONDITIONS: Cervical Disease
Keywords: Spectroscopy; HPV
MeSH Terms: conditions — Uterine Cervical Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — cells from the cervix to collect and test for HPV
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Negative and Referral Cytology Results: CNDS Advanced Cervical Scan Colposcopy
  Interventions: Device: CNDS Advanced Cervical Scan

INTERVENTIONS:
Device: CNDS Advanced Cervical Scan — Subjects (approximately 500) will be initially enrolled from a general screening population in the first phase, and during the second phase from the colposcopy clinic population (approximately 300) based on their referral abnormal Pap cytology conducted within 120-days in order to achieve a statistically viable number of normal women, women with CIN1/2 and women with CIN3+, as described in Section 6.1, "Cervical Cytology Enrollment Targets". After the CNDS test, a sample for Hybrid Capture 2 HPV testing and liquid cytology will be collected in addition to colposcopy and biopsy, if indicated.

SUMMARY:
The purpose of this study is to evaluate whether fluorescence and reflectance spectroscopy can improve the ability to detect the presence of premalignant lesions on the cervix.

DETAILED DESCRIPTION:
Subjects (approximately 500) will be initially enrolled from a general screening population in the first phase, and during the second phase from the colposcopy clinic population (approximately 300) based on their referral abnormal Pap cytology conducted within 120-days in order to achieve a statistically viable number of normal women, women with Cervical Intra-epithelial Neoplasia (CIN1/2) and women with CIN3+, as described in Section 6.1, "Cervical Cytology Enrollment Targets". After the Cervical Neoplasia Detection System (CNDS) test, a sample for Hybrid Capture 2 Human papillomavirus (HPV) testing and liquid cytology will be collected in addition to colposcopy and biopsy, if indicated.

A key component of effective screening studies designed to evaluate new detection modalities is verification of the gold standard comparison by which estimates of sensitivity and specificity are generated. In the case of screening studies in general and studies of cervical disease detection in particular, the avoidance of verification bias is a priority. For the purposes of the proposed study, CIN3 or cancer (CIN3+) must be verified or adjudicated by multiple histopathologists. Results for women with CIN1 or CIN2 will be confirmed histopathologically and analyzed as a separate subgroup because these lesions often regress to normal in certain populations and tend to cause disagreement among histopathologists. In order to verify absence of disease (i.e., CIN1 or less severe), the investigators will not rely on histopathology, as it would not be ethical to perform multiple biopsies or excisional procedures to obtain a tissue sample for histopathology. Instead, women will be considered normal if they have negative referral cytology, are free of high risk HPV and are colposcopically normal.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 or above
* Able to read or understand and give informed consent
* Negative pregnancy test or documentation of acceptable birth control
* Willing to undergo colposcopy, cytology (if required) and HPV testing on day of study
* Abnormal cytology result within 120 days of CNDS test for Phase 2 subjects

Exclusion Criteria:

* Pregnancy
* Menstruating
* Previous cervical neoplasia
* Prior hysterectomy
* Conditions relating to the cervix that would render the test difficult to perform, including but not limited to:

Excessive blood or mucus that cannot be removed Abnormal congenital cervix Unable to tolerate speculum or CNDS single use cervical guide

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: General screening population Scheduled for colposcopy
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2014-08; Primary Completion 2015-09 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy including sensitivity, specificity and predictive values | for each participant approximately 30 days to collect data, no follow up data collected
  Collect clinical data for re-calibrating the processing of spectral data from the CNDS for eventual use as a primary screening modality. Resampling or other cross validation methods will be used to estimate the sensitivity, specificity and predictive values of a screening algorithm based on the recalibrated spectral data. These estimates will be used to compare with those of existing screening and diagnostic modalities such as Pap based cytopathology, HPV DNA testing and/or VIA (Visual Inspection with Acetic Acid).

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 30 days, no follow up inteneded
  Is the CNDS safe when used as directed and that the test procedure is accepted by both physicians and their patients.

CONTACTS AND LOCATIONS:
Overall Officials: Daron G Ferris, MD, Principal Investigator — Augusta University
Locations (1):
- Georgia Regents University, Augusta, Georgia, United States

REFERENCES:
- [Result] Twiggs LB, Chakhtoura NA, Ferris DG, Flowers LC, Winter ML, Sternfeld DR, Lashgari M, Burnett AF, Raab SS, Wilkinson EJ. Multimodal hyperspectroscopy as a triage test for cervical neoplasia: pivotal clinical trial results. Gynecol Oncol. 2013 Jul;130(1):147-51. doi: 10.1016/j.ygyno.2013.04.012. Epub 2013 Apr 13. PMID 23591399